CLINICAL TRIAL: NCT00164567
Title: IPV Screening in Health Care Clinics in Rural South Carolina
Brief Title: Intimate Partner Violence (IPV)Screening in Health Care Clinics in Rural South Carolina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of South Carolina (Other); The University of Texas Health Science Center, Houston (Other); University of North Carolina, Chapel Hill (Other); Pee Dee Coalition (Other); Care South, Inc. (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3142; US4/CCU419014
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Partner Abuse
Keywords: partner abuse; screening; intimate partner violence

INTERVENTIONS:
Behavioral: Onsite IPV specialist
Behavioral: Empowerment focused intervention

SUMMARY:
The purpose of this study is to implement universal screening for intimate partner violence (IPV) and to test two clinic-based interventions for women who screen positive for current or recent IPV. The study population will be implemented in Pee Dee region of the state of South Carolina and will include primarily low-income women who seek care at selected primary health care clinics in the region.

In this study, all women 18 and older receiving care at selected primary care clinics will be offered screening for IPV annually. Clinicians will use a structured screening tool to assess physical, sexual, and psychological IPV in a current relationship (IPV+) or IPV experienced by the woman in the past five years (Recent IPV). Clinics will be randomly assigned to implement a clinic-based intervention for women who screen positive for current or recent IPV. Two interventions will be implemented using a factorial design. In the Empowerment-Focused Patient Education Intervention, clinicians will conduct a 7-session intervention focusing on the health and well-being of the woman and attempt to link women's IPV experience with their health. In the IPV Services Intervention, IPV Specialists who are trained advocates from the Pee Dee Coalition Against Domestic and Sexual Assault (PDC) will be based in the clinic to (a) counsel women about IPV including safety planning, (b) provide linkages to PDC services, and (c) link women to clinic-based support groups developed specifically for this project.

We hypothesize the intervention(s) will change (a) clinician screening, referral, and IPV documentation patterns, (b) clinician IPV knowledge and perceived skills in working with women who have experienced IPV and their children (c) women's help-seeking behaviors, risk of poor mental and physical health, and (d) women's risk of subsequent IPV victimization. To evaluate these outcomes, we will survey clinicians and prospectively follow a group of consenting IPV+ women (N=300 in each intervention arm) to assess changes in their help-seeking, health behavior and status, IPV experience over two-years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 - 65 years
* must screen positive for partner abuse

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200

PRIMARY OUTCOMES:
help-seeking
physical health
Psychological health

SECONDARY OUTCOMES:
revictimization from partner violence
child behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Ann Coker, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Care South clinics (Various), Hartsville, South Carolina, United States